

(Protocol Synopsis)

| 文件編碼 | KMUH/IRB/SOP/02.01.O |
|------|----------------------|
| 版次 | 2024.00 |

| I. | Protocol title: Effects of an Exercise Snack Intervention on Employee Health and Work |
|---|---|
| Perf | formance: A Study at Kaohsiung Medical University |
| п. | Objectives: |
| (1) | To develop brief exercise videos targeting different areas of physical discomfort (e.g., neck |
| | and shoulders, lower back, lower limbs), specific fitness goals (e.g., localized muscle |
| | stretching, targeted muscle strengthening, cardiorespiratory endurance, balance training), |
| | high-intensity interval training (HIIT), or the acquisition of specific movement skills (e.g., |
| | core stability, pelvic floor muscle contraction, and multi-directional pelvic mobility). |
| (2) | To design personalized exercise "menus" based on individual needs identified through a |
| | preliminary assessment, with the goal of improving adherence to voluntary exercise routines |
| | among staff. |
| (3) | To apply the concept of "exercise snacking" by implementing a daily routine of 3 to 8 brief |
| | exercise sessions, and to evaluate changes in staff members' physiological health, work |
| | performance, and exercise behavior after a 12-week intervention. |
| Ш. | Test drug |
| 1. | Name: Not applicable |
| 2. | Dosage form: Not applicable |
| 3. | Dose(s): Not applicable |
| 4. | Dosing schedule: Not applicable |
| 5. | Mechanism of action: Not applicable |
| 6. | Pharmacological category: Not applicable |
| IV. | Study design |
| 1. | ☐ Control: ☐ placebo |
| | ☐ active (please specify name and dosage) |
| | □ others |
| | ■ Uncontrolled |
| 2. | Blinding: ■ open-label □ single blind □ double blind □ others |
| 3. | Randomized: ☐ yes ■ no |
| 4. | ■ Parallel □ cross-over □ others |
| 5. | Sample/Data |
| | $\square$ Biospecimens(IF sourced from the biological database $\square$ No $\square$ Yes, Name:) |
| | □Excluding DNA extraction |
| | □Including DNA extraction |

1



(Protocol Synopsis)

| 文件編碼 | KMUH/IRB/SOP/02.01.O |
|------|----------------------|
| 版次 | 2024.00 |

| | | edical record data |
|---|---|---|
| | Q | uestionnaires |
| | R | ecord (including measurements, interviews, voice recordings, video |
| | rec | ordings |
| | □В | ig data |
| | <u></u> 0. | thers: |
| 6. | Dura | ation of study: from IRB approval ~to 12, 31, 2028, total 43 months |
| | Dura | ation of Enrollment: from IRB approval ~to 12, 31, 2028, total 43 months |
| Dura | atio | n of treatment: from IRB approval ~to 12, 31, 2028, total 43 months |
| | Dura | ation of follow-up: from IRB approval ~to 12,31,2028, total 43 months s |
| 7. | | Multi-national □multi-center(Taiwan) ■single center(Taiwan) |
| 8. | Numl | per of subjects: |
| 9. | Is · | there any of the followings included DSMB, Data Safety Monitoring Board: |
| | | yes ■ no |
| <b>V</b> | Asse | ssment criteria |
| 1. | . Efficacy: Physical fitness assessments, Performance on functional movement tasks | |
| 2. | Saf | ety: Not applicable |
| 3. | Pha | rmacokinetics: Not applicable |
| 4. | Qua | lity of life: Perceived stress scale, Work performance, Burnout inventory |
| VI. | Sel | ection criteria |
| 1. | Mai | n inclusion criteria: |
| | (1) | Currently employed at Kaohsiung Medical University or Kaohsiung Medical University |
| | | Hospital. |
| | (2) | Willing to participate in a 12-week exercise intervention, complete related |
| | | questionnaires, and undergo physical performance assessments. |
| 2. | Mai | n exclusion criteria: |
| | (1) | Pregnant individuals, due to safety concerns related to exercise intensity and physical |
| | | assessments. |
| | (2) | Individuals with a diagnosed neurological disorder (e.g., stroke, Parkinson's disease). |
| | (3) | Individuals experiencing severe pain in the upper or lower limb joints that interferes |
| | | with their ability to complete the assessments. |
| | (4) | Individuals assigned to high-intensity exercise who have unstable cardiac conditions |
| | | (e.g., angina, myocardial infarction, heart failure). |



(Protocol Synopsis)

| 文件編碼 | KMUH/IRB/SOP/02.01.O |
|------|----------------------|
| 版次 | 2024.00 |

#### VII. Study procedures(summary)

- 1. Written informed consent must be obtained before any study specific procedures are undertaken.
  - (1) Recruitment announcements will be distributed through internal communication channels at Kaohsiung Medical University and its affiliated hospital.
  - (2) An introductory session and practical workshop on the "exercise snacking" program will be held.
  - (3) Participants will complete the informed consent form and attend a brief interview to complete questionnaires, including basic information (e.g., exercise habits) and a "personal issues and exercise needs assessment" to assist in designing a personalized exercise menu.

#### 2. The process of the experiment (brief describe)

- (1) Pre-intervention assessment: Participants will undergo baseline testing within one week prior to the start of the exercise intervention.
- (2) Intervention period: Participants will engage in a 12-week exercise intervention program.
- (3) Post-intervention assessment: Within one week following the intervention, participants will complete follow-up assessments.
- (4) Follow-up check: One month after the completion of the program, participants will be contacted to assess whether they have continued engaging in the exercises independently without supervision from the research team.

#### VIII. Concomitant treatment:

1. Permitted: Not applicable

2. Prohibited: Not applicable

#### IX. Statistical analysis

#### 1. Statistical Method for Efficacy / Safety measurements:

This study adopts a cross-sectional data collection approach, and all data analyses will be conducted using SPSS version 20. The normality of continuous variables will be assessed using the One-Sample Kolmogorov–Smirnov test. Based on the results of the normality test, appropriate statistical methods will be selected.

If the data are normally distributed, parametric tests such as the paired-sample t-test will be used to compare pre- and post-intervention differences. If the data are not normally distributed, non-parametric tests such as the Wilcoxon signed-rank test will be employed.

Additionally, correlations between variables will be analyzed using either Pearson's correlation



(Protocol Synopsis)

| 文件編碼 | KMUH/IRB/SOP/02.01.O |
|------|----------------------|
| 版次 | 2024.00 |

coefficient (for normally distributed data) or Spearman's rank correlation coefficient (for non-normally distributed data).

4 Version: Version 1 Date:05/15/2025